CLINICAL TRIAL: NCT04136743
Title: Ultrasound-Guided Treatments for Chronic Shoulder Pain in Wheelchair Users With Spinal Cord Injury: A Randomized Controlled Trial
Brief Title: Ultrasound-Guided Treatments for Shoulder Pain in Wheelchair Users With Spinal Cord Injury
Acronym: MFAT-SCI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-1066-19
Record Dates: First submitted 2019-07-01; First posted 2019-10-23 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Spinal Cord Injuries; Tendinopathy; Rotator Cuff Tears; Shoulder Pain
Keywords: Rehabilitation; Regenerative Medicine; Regenerative Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Tendinopathy; Rotator Cuff Injuries; Shoulder Pain | interventions — Dexamethasone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor will be blinded to treatment group when analyzing data for publication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Corticosteroid (Active Comparator): Participants will receive a corticosteroid injection (BMS, Kenacort-A 40 mg [triamcinolone acetonide]) into the subacromial space under direct ultrasound guidance by means of a 5-mL syringe with a 22-guage needle.
  Interventions: Drug: Dexamethasone
- Micro-Fragmented Adipose Tissue (Experimental): Participants will receive a single injection of micro-fragmented adipose tissue into the lesion (e.g. tear, subacromial bursa, glenohumeral joint, acromioclavicular joint) under ultrasound guidance using an 18 gauge x 3.5 inch needle.
  Interventions: Device: Lipogems

INTERVENTIONS:
Device: Lipogems — The Lipogems system (Lipogems International SpA, Milan, Italy) is designed to isolate autologous, micro-fragmented adipose tissue without enzymes or other additives. It uses mild mechanical forces to break down adipose tissue that is extracted from the patient into a form that can be injected into the tendon lesion and other degenerated tissues in a sterile and safe manner. The resulting product is rich in pericytes and mesenchymal stromal cells, retained within an intact stromal vascular niche, that is ready for use in clinical applications.
  Other Names: Micro-fragmented Adipose Tissue
  Arms: Micro-Fragmented Adipose Tissue
Drug: Dexamethasone — Triamcinolone Acetonide is a corticosteroid, which is a class of drugs that are commonly prescribed for shoulder pain. They work to reduce pain by limiting inflammation. They are typically injected into the subacromial space with or without ultrasound guidance.
  Other Names: Corticosteroid
  Arms: Corticosteroid

SUMMARY:
Rotator cuff disease (i.e., rotator cuff tendinopathy or tear) is a common cause of shoulder pain in persons with chronic spinal cord injury (SCI). It usually resolves with non-operative treatments such as pharmacological agents and physical therapy; however, when this fails, rotator cuff surgery may be the only option. Corticosteroid injections are another alternative to provide temporary relief, but can over time accelerate degeneration of the tendon and lead to further damage. Autologous adipose tissue injection has recently emerged as a promising new treatment for joint pain and soft tissue injury. Adipose can be used to provide cushioning and filling of structural defects and has been shown to have an abundance of bioactive elements and regenerative perivascular cells (pericytes). The purpose of this study is to explore the efficacy of autologous, micro-fragmented adipose tissue (Lipogems®) injection under ultrasound guidance for chronic shoulder pain in persons with SCI compared with the standard-of-care, corticosteroid injection.

DETAILED DESCRIPTION:
This is randomized controlled trial to determine the efficacy of autologous, micro-fragmented adipose tissue (MFAT) injection under ultrasound guidance for chronic, nonresponsive shoulder pain due to rotator cuff disease (i.e., rotator cuff tendinopathy) in persons with spinal cord injury (SCI). The control for this study, to which MFAT will be compared, is corticosteroid injection into the subacromial space. Twenty-four (24) persons with SCI who have chronic shoulder pain for longer than 6 months in spite of completing conservative treatment and who are diagnosed with rotator cuff disease on examination will be recruited.

MFAT Group: Micro-fragmented adipose tissue will be obtained by using a minimal manipulation technique in a closed system (Lipogems®), without the addition of enzymes or any additives. The final product will consist of micronized fat tissue yielding fat clusters with preserved vascular stroma of about 500 microns with intact stromal vascular niches and harboring regenerative cellular elements. Approximately 6 mL of micro-fragmented adipose will be injected into the tendon with a 22-gauge needle under continuous ultrasound guidance. No other biological or pharmacological agents will be used in combination with the micro-fragmented adipose.

Corticosteroid Group: In the corticosteroid group, participants will receive a corticosteroid injection (BMS, Kenacort-A 40 mg [triamcinolone acetonide]) into the subacromial space under direct ultrasound guidance by means of a 5-mL syringe with a 22-guage needle.

Both Groups: After 24 hours, participants will be given a standardized stretching protocol to follow for 4 weeks followed by a formal strengthening program. Participants will be followed for adverse events and changes in shoulder pain intensity on an 11-point numerical rating scale (NRS; 0-10, with anchors "no pain" and "pain as bad as you can imagine"); the Wheelchair User's Shoulder Pain Index (WUSPI; 15-item disease-specific functional measure of shoulder pain in persons with SCI); the PROMIS Physical Functioning short form; the Brief Pain Inventory interference items (BPI-I7; a subscale of 7 items measuring interference with general activity, sleep, mood, relationships, etc.); and a 5-point subject global impression of change (SGIC) scale. Subjects will be examined at 1 month, 2 months, 3 months, and 6 months after the treatment. In addition to subjective outcome measures, quantitative ultrasounds will be conducted at baseline, 1 month, 2 months, 3 months, and 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 to 70 years of age, inclusive
* Neurological impairment secondary to a spinal cord injury or disorder that occurred at least twelve (12) months prior to the Screening Visit and the level of the injury is between C6 and L5, inclusive
* Non-ambulatory except for exercise purposes and uses a manual or power wheelchair as his/her primary means of mobility (> 40 hours/week)
* Currently has chronic shoulder pain due to rotator cuff disease in spite of at least 6 months of conservative treatment
* Average shoulder pain intensity during the week leading up to the Screening Visit is at least 4 out of 10 on an 11-point numerical rating scale (NRS; 0, no pain; 10, maximum pain imaginable).
* Rotator cuff disease will be defined as pain over the anterior shoulder, with direct palpation and pain at the shoulder with provocative tests for rotator cuff disease that is confirmed by tendinopathic changes on ultrasound imaging.

Exclusion Criteria:

* Report prior MFAT treatment
* Have a history of systemic disorders, such as diabetes or rheumatoid arthritis
* Have a contra-indication to the procedure, such as infection, coagulopathy, or currently taking anti-coagulant
* Report having a glucocorticoid injection in the past 4 weeks
* Are pregnant
* Have any medical condition, including psychiatric disease, which would interfere with the interpretation of the study results or the conduct of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-06-14 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Numerical Rating Scale | 6 months
  Shoulder pain intensity will be assessed using an 11-point numerical rating scale (NRS; 0-10, ranging from 0 = "no pain" to a maximum of 10= "pain as bad as you can imagine". Pain intensity is the most common pain domain assessed in research and clinical settings. Although different rating scales have proven to be valid for assessing pain intensity, the 11-point NRS has the most strengths and fewest weaknesses of available measures. An 11-point NRS measure of pain intensity allows for comparison across clinical trials of chronic pain treatment and has been recommended by the IMMPACT consensus group for use in pain clinical trials and by the 2006 NIDRR SCI Pain outcome measures consensus group. We will evaluate changes in scores between baseline and 6 months.

SECONDARY OUTCOMES:
Wheelchair User's Shoulder Pain Index | 6 months
  Activity-dependent shoulder pain intensity will be assessed using the Wheelchair Users Shoulder Pain Index (WUSPI). The WUSPI is a 15-item self-report instrument that measures shoulder pain intensity in wheelchair users during various ADLs over the past week; for example, transfers, loading a wheelchair into a car, wheelchair mobility, dressing, bathing, overhead lifting, driving, performing household chores, and sleeping. Each item is scored using a 10cm visual analog scale (VAS) which is anchored at the ends with "no pain" and "worst pain ever experienced." Individual item scores are summed to arrive at a total index score, which ranges from 0 to 150. We will evaluate changes in scores between baseline and 6 months.
Patient Global Impression of Change | 6 months
  The subject will be asked to rate on a 7-point scale his or her overall impression following treatment as compared to the previous measurement interval. The 7-point PGIC scale (also referred to as the original Guy/Farrar-PGIC scale; anchored by "very much improved" and "very much worse") is used to measure global treatment effect and is recommended as a compliment to unidimensional pain intensity scales. Although other versions of the PGIC scale exist, the SCI Measures Pain Committee recommends using the original Guy/Farrar-PGIC scale in clinical trials since it has been used extensively and been shown to be sensitive to change. We will evaluate scores at 6 months.
Physical Examination of the Shoulder Scale | 6 months
  The PESS will be derived from findings during the shoulder examination performed. The PESS was developed to apply a grading system to commonly-used provocative tests for the diagnosis of shoulder soft-tissue disorders. Eleven physical examination maneuvers are given a score dependent upon the pain elicited: 0 (no pain), 1 (equivocal for pain), or 2 (pain present). The scores are summed for a total between 0 and 22. The physical examination maneuvers include: biceps tendon/bicipital groove tenderness; supraspinatus tendon/greater tuberosity tenderness; acromioclavicular joint tenderness; resisted external rotation; resisted internal rotation; supraspinatus test; painful arc test; Neer impingement sign; Hawkins-Kennedy impingement sign; O'Brien active compression test for acromioclavicular joint and labral pathology. We will evaluate changes in scores between baseline and 6 months.
Ultrasound Shoulder Pathology Rating Scale | 6 months
  All participants will undergo a clinical ultrasound examination. The ultrasound will be performed by a physiatrist with musculoskeletal ultrasound training. The Ultrasound Shoulder Pathology Rating Scale (USPRS) applies a grade to seven ultrasound findings for shoulder pathology. The scale is designed to give an impression of global shoulder pathology associated with overuse. A score of 0 indicates no observable pathology, up to a maximum of 23. The exams include biceps tendinosis/tendinopathy; supraspinatus tendinosis/tendinopathy; greater tuberosity cortical surface irregularities; bursal thickening; joint edema; dynamic supraspinatus and subscapularis impingement. We will evaluate changes in scores between baseline and 6 months.
Quantitative Ultrasound of the Supraspinatus Tendon | 6 months
  Quantitative ultrasound protocols will be used to evaluate changes in morphological and structural characteristics of the supraspinatus tendon after treatment. We will collect conventional B-mode ultrasound images alongside shear wave elastography images and apply custom image analysis algorithms to quantify the parameters of interest. Greyscale parameters of interest include tendon thickness and mean echogenicity (i.e. "brightness"), which are reflective of inflammation and edema. This method will be adapted based on a previously-validated technique that has been used in wheelchair users with SCI. The primary elastography parameter of interest is strain ratio; that is, the strain within the ROI relative to a reference point in the deltoid muscle immediately outside the tendon. We will evaluate changes in greyscale and shear wave parameters between baseline and 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

REFERENCES:
- [Background] Cherian C, Malanga GA, Hogaboom N, Pollack MA, Dyson-Hudson TA. Autologous, micro-fragmented adipose tissue as a treatment for chronic shoulder pain in a wheelchair using individual with spinal cord injury: a case report. Spinal Cord Ser Cases. 2019 May 13;5:46. doi: 10.1038/s41394-019-0186-8. eCollection 2019. PMID 31632705
- [Background] Randelli P, Menon A, Ragone V, Creo P, Bergante S, Randelli F, De Girolamo L, Alfieri Montrasio U, Banfi G, Cabitza P, Tettamanti G, Anastasia L. Lipogems Product Treatment Increases the Proliferation Rate of Human Tendon Stem Cells without Affecting Their Stemness and Differentiation Capability. Stem Cells Int. 2016;2016:4373410. doi: 10.1155/2016/4373410. Epub 2016 Jan 6. PMID 27057170